CLINICAL TRIAL: NCT03614910
Title: Ablation of Unresectable Locally Advanced Pancreatic Cancer With Nanoknife Irreversible Electroporation (IRE) System: Response and Tolerability
Brief Title: Ablation of Unresectable Locally Advanced Pancreatic Cancer With Irreversible Electroporation (IRE) System
Status: Completed | Type: Observational
Sponsor: Holy Name Medical Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: holynamenanoknife1
Record Dates: First submitted 2018-07-12; First posted 2018-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced pancreatic cancer; irreversible electroporation; Nanoknife
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Locally Advanced Pancreatic Cancer: Patients with locally advanced unresectable pancreatic cancer. Unresectable tumors as defined by:
  * occlusion, thrombosis or several centimeters of encasement of the superior mesenteric vein or portal vein
  * tumor abutment greater than 180 degrees of the superior mesenteric artery or thrombosis of the artery
  * abutment or encasement of the celiac axis
  * involvement of lymph nodes outside the area of resection
  Interventions: Device: Nanoknife Irreversible Electroporation

INTERVENTIONS:
Device: Nanoknife Irreversible Electroporation — Irreversible electroporation will be delivered between electrodes that are placed by intraoperative ultrasound guidance around the tumor

SUMMARY:
Patients with pancreatic ductal adenocarcinoma will be screened by pancreatic protocol cross-sectional imaging to see if they have locally advanced unresectable pancreatic ductal adenocarcinoma. Patients with unresectable disease will undergo at least four cycles of standard of care chemotherapy before being re-evaluated for treatment with irreversibe electroporation (i.e., Nanoknife). If patients are over 18 years of age, have pancreatic tumor size less than 5cm, and can safely undergo a laparotomy, they will be considered for participation. The patient cannot undergo the procedure if they have metastatic disease, a pacemaker or an electrostimulator, a metallic stent that cannot be exchanged, a convulsive (i.e., epilepsy) condition, an estimated survival less than three months, atrial fibrillation with an undetectable waveform on ECG sync device, severe cardiac disease, a international normalised ratio (INR) that is less than 1.5, or a performance status >2.

For the procedure, a laparotomy will be performed and Nanoknife probe placement will be done under intraoperative ultrasound. The number of probes, depth of the probes and rapid pulse series will be decided by the surgeon and are based on the size and location of the desired area of ablation.

Patients will be followed for overall survival, progression-free survival, tumor response, tumor markers, symptom improvement, and complications. Symptom improvement will be measured by assessment of pain, quality of life, total bilirubin if biliary obstruction is initially present, and oral intake if gastric outlet obstruction is initially present. They will have regular follow up with the surgeon that will include routine surveillance imaging and blood work.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma is extremely aggressive and is the 4th most frequent tumor-related cause of death in the Western world. The one-year survival rate is 20 percent and the 5-year overall survival rate is only 5 percent. Pancreatic ductal adenocarcinoma often become symptomatic at very advanced stages with only 15 to 20 percent of patients being able to undergo a therapeutic local resection. Patients who do not meet the criteria for local consolidative resection may either have advanced locoregional disease and/or distant metastases. Advanced locoregional pancreatic ductal adenocarcinoma without metastatic disease has a survival rate of 6 to 12 months. Those with distant metastases have a survival rate of only 3 to 6 months.

Locally advanced pancreatic adenocarcinoma is defined by the involvement of the superior mesenteric artery, the celiac axis, and/or long segment portal vein occlusion on cross-sectional imaging. Resectable tumors will be free from the superior mesenteric vein, superior mesenteric artery and celiac axis, with no nodal involvement outside of the area of resection. Unresectable disease will have occlusion, thrombosis or encasement that extends for several centimeters of superior mesenteric vein and portal vein. Tumor abutment, encasement or thrombosis of the superior mesenteric artery is also considered unresectable disease. Involvement of lymph nodes outside of the area of resection also indicates that the patient is not resectable.

For patients who have unresectable pancreatic ductal adenocarcinoma, chemotherapy and radiation can only provide short-term disease control. Chemotherapy and radiation regimens have not been shown to prolong survival significantly in this disease, and therefore, there is a need for additional adjunctive or consolidative treatment to provide improved local control, pain relief and possibly impact survival. Image guided ablation technique like irreversible electroporation has shown promise as a new treatment option for patients with stage III locally advanced pancreatic cancer.

A unique advantage of Nanoknife is that it does not require heat to ablate tumor cells, rather it works by using high voltage but low energy direct current. The process in which low energy direct current ablates tissue is called irreversible electroporation. In order to understand how this process works, the investigators have to understand some background cell biology. The cell membrane separates the intracellular space and the extracellular space/fluid, and controls transport processes between the two compartments of the cell. Electroporation increases cell membrane permeability by subjecting it to an electrical field and uses rapid series of short electrical pulses delivered using high voltage but low energy direct current to create defects (pores) in the cell membrane that result in loss of homeostasis and cell death. The result is a well demarcated area of ablation. The Nanoknife system comes with 19 gauge needles that have depth markings. The needle surface is echogenic. The active electrode length is adjustable in 0.5 cm increments from zero to 4 cm. There is an external electrocardiogram synchronization device that automatically detects the R wave and energy is delivered synchronously to the R wave. The electrodes can be arranged in multiple configurations using two to six electrodes. The spacing between the electrodes can be from 0.5 cm to 2.0 cm, and electrode exposure can be from 0.5 cm to 4.0 cm. Energy is delivered between the electrode pairs, and this results in an area of ablated tissue.

Nanoknife is particularly useful in patients with pancreatic ductal adenocarcinoma because of the proximity of pancreatic tumors to critical surrounding structures such as bile ducts and major blood vessels. Because it does not use heat to ablate tissue (which induces necrosis) but rather uses cell apoptosis, it theoretically has no impact on the surrounding structures that mainly consist of proteins like vascular elastic and collagenous structures as well as peri-cellular matrix proteins (protecting large blood vessels and bile ducts). Further study of Nanoknife is needed to see if this therapy can potentially impact survival and/or provide adequate local palliation to improve quality of life in patients with locally advanced unresectable pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* locally advanced unresectable pancreatic ductal adenocarcinoma as demonstrated by CT or MRI
* must have received standard chemotherapy and completed at least four cycles of treatment at least 5 weeks prior to therapy with Nanoknife
* INR <1.5
* able to tolerate laparotomy (medical/cardiac clearance as needed)
* able to comply with protocol requirements
* women of childbearing potential must have a negative serum pregnancy test and be practicing an effective form of birth control

Exclusion Criteria:

* patients with tumor >5cm after completion of chemotherapy
* presence of metastatic disease
* patients with a pacemaker or electrostimulator
* estimated survival is less than 3 months
* presence of a metallic stent (biliary or duodenal) which cannot be removed or exchanged for plastic
* ECOG performance status more than or equal to 2
* epilepsy or other convulsive conditions
* cannot tolerate general anesthesia
* patients with atrial fibrillation who have an undetectable wave form on the ECG synchronization device
* patients with inducible ischemia on cardiac stress test or uncontrolled angina
* white blood cell count less than or equal to 2,000, absolute neutrophil count <1,000, platelets <50,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced unresectable pancreatic cancer who meet the criteria for Nanoknife and are able to safely undergo a laparotomy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 10 years
  Time from Nanoknife treatment to the patient's death
Local progression-free survival | up to 10 years
  Time from Nanoknife treatment to local disease progression
Distant disease-free survival | up to 10 years
  Time from Nanoknife treatment until distant disease development
Tumor response | First year
  Change in tumor size in response to Nanoknife treatment using RECIST criteria V1.1 (CR, PR, SD, PD)

SECONDARY OUTCOMES:
Complications | 90 days
  The incidence of the following complications after treatment with Nanoknife will be recorded: hematologic, ileus, bile leak, portal vein thrombosis, deep vein thrombosis, pulmonary, renal failure, ascites, wound infection, dehydration/failure to thrive/nausea, bleeding, diarrhea, duodenal leak, liver insufficiency, pancreatic leak
Tumor Markers | up to 10 years
  CA 19-9 will be measured at 6 weeks post op, 3 months post op, 6 months post op, 1 year post op, then yearly
Biliary Obstruction | up to 10 years
  Change in biliary obstruction after treatment will be recorded using total bilirubin and conjugated/unconjugated bilirubin levels at each follow up office visit
Gastric outlet obstruction | up to 10 years
  Gastric outlet obstruction after treatment will be monitored with symptoms resulting in decreased oral intake (nausea, vomiting, and inability to eat). Objectively we will also measure patient weight in kilograms at each office visit.
Cancer related pain | up to 10 years
  Cancer related pain after treatment will be measured using Visual Analog Pain scale 0-10, zero being no pain and 10 being worst pain possible. Pain scale will be assessed at each follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Kwon, MD, Principal Investigator — Holy Name Medical center
Locations (1):
- Holy Name Medical Center, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No